CLINICAL TRIAL: NCT03108521
Title: Study on Polymorphism of DPP-4 and GLP-1R Genes in Chinese Population and Its Empirical Study on Treatment of Diabetes
Brief Title: SNP Study of DPP-4 and GLP-1R in Chinese People (Including Diabetes Patients)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Enwu Long, Chief Pharmacist, Sichuan Provincial People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015SZ0182
Record Dates: First submitted 2017-01-04; First posted 2017-04-11 (Actual); Results first posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus
Keywords: DPP-4; GLP1R ; gene polymorphism research; diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin group (Experimental): Patients in this group will accept Sitagliptin phosphate tablets as their intervention. Specifications: Each tablet 100mg (with sitagliptin dollars). Regimen: The recommended dose is 100mg.QD for 3 months.
  Interventions: Drug: Sitagliptin
- non-T2DM group (No Intervention): Subjects in this group are T2D free. We use their gene information to study SNP differences between T2D patients and non-T2DM people.

INTERVENTIONS:
Drug: Sitagliptin — 100mg.QD for 3 months
  Other Names: Januvia
  Arms: Sitagliptin group

SUMMARY:
Incretin-based therapy is currently one of the most popular diabetes treatment approaches. However, differences of response ware found in previous studies. We hypothesis that SNPs of DPP-4, GLP-1 and GLP-1R genes may play crucial roles in the response differences. Therefore, this study aims to investigate the correlation of incretin-related gene polymorphism and individual differences in the response of DPP-4 inhibators (take Sitagliptin as an example). In addition, The distribution differences of the SNPs in diabetics and non-diabetics are evaluated to study the relationships between the SNPs and diabetes onsets.

DETAILED DESCRIPTION:
Single Nucleotide Polymorphism (SNP) plays an important role in the differences of clinical manifestations and drug responses of diseases. The vast majority of SNP sites are located in the non-coding region of the gene (about 95%), which is called SNP(non-coding SNP (ncSNP), while the other part of SNP is located in the coding region of the gene, which is called coding SNP (cSNP). Furthermore, cSNP can be divided into two categories: SNP that does not change the encoded amino acid sequence is called synonymous SNP(synonymous SNP, SSNP); SNP that changes amino acid sequence is called SNP(non-synonymous SNP (NSNP). Although not involved in coding amino acid, some ncSNPs may also affect the regulation of protein expression. Therefore, it is of great significance to study the effects of NC SNP and cSNP on the occurrence and development of diseases and drugs.

DPP-4 enzyme inhibitor is combined with DPP-4 enzyme in human body to reduce hydrolysis of active GLP-1, thus increasing the level of endogenous active GLP-1. Active GLP-1 combines with its receptor GLP-1R to promote insulin release and inhibit glucagon release in hyperglycemia state, and produces opposite effect in hypoglycemia state.

Based on the above principles, we speculate that SNP of genes that may affect the hypoglycemic effect of DPP-4 enzyme inhibitor are:

1. SNP of DPP-4 enzyme gene. SNP of DPP-4 enzyme gene may affect the enzyme activity and/or protein expression level of DPP-4. Assuming that the effect of DPP-4 enzyme inhibitor is sufficient, patients with higher DPP-4 enzyme activity are more sensitive to DPP-4 enzyme inhibitor drugs; However, for patients with low DPP-4 enzyme activity, DPP-4 enzyme inhibitor drugs cannot play a stronger role in lowering blood sugar.
2. SNP of GLP-1 gene. SNP of GLP-1 gene may affect activity or expression level of GLP-1. Patients with high GLP-1 level are more sensitive to DPP-4 enzyme inhibitor drugs.
3. SNP of GLP-1R gene. SNP of GLP-1R gene may affect activity or expression level of GLP-1R. Patients with high GLP-1R level are also more susceptible to DPP-4 enzyme inhibitor drugs.

However, studies on the hypoglycemic effect of DPP-4, GLP-1 and their receptors on DPP-4 enzyme inhibitors in the treatment of T2DM are rare, which is not conducive to the evaluation of individualized treatment of such drugs. Therefore, this chapter intends to select SNP sites with high mutation frequencies of DPP-4, GLP-1 and GLP-1R genes to study the mutation frequencies of these SNPs in diabetic patients and non-diabetic patients and their effects on DPP-4 enzyme inhibitor sitagliptin's hypoglycemic effect on T2DM patients.

ELIGIBILITY:
For Sitagliptin group--

Inclusion Criteria:

1. According to diagnostic criteria from Chinese type 2 diabetes prevention and treatment guidelines in diabetes, that published in the Chinese Medical Association Diabetes credits in 2010: Symptoms of diabetes (polydipsia, polyphagia, polyuria, weight loss, itchy skin, blurred vision and other acute metabolic disorders performance caused by hyperglycemia) and RBG≥11.1mmol/L, or fasting plasma glucose (FPG)≥7.0mmol/L, or plasma glucose of 2 hours post glucose-load≥11.1 and patients diagnosed with type 2 diabetes; HbA1c in the range of 7%-10%;
2. Age 40-70 years;
3. Body Mass Index(BMI) 18-40;
4. Did not accepted any antihyperglycemic therapies during the past 4 weeks, or did not change their antihyperglycemic treatment plan in the past 3 months;
5. Did not participate in clinical trials within three months;
6. No serious heart, brain, liver and kidney disease;
7. Signed informed consent.

Exclusion Criteria:

1. Have taken any incretin drugs within recent 1 month;
2. Patients with a weakened immune system;
3. C-peptide < 0.3ng/ml;
4. GLP-1 and DPP4-i drugs allergies;
5. Pregnancy and breast-feeding patients;
6. Patients taking drugs that may affect the metabolism of GLP-1 and DPP4;
7. Patients have serious heart, liver, kidney and respiratory dysfunction; Patients have medullary thyroid carcinoma (MTC) with past history or family history, as well as multiple endocrine neoplasia type 2 syndrome (MEN2);
8. Drug abusing and alcoholism within a year.

For non-T2D group--

No major diseases such as tumors, no dyslipidemia, chronic diseases such as hypertension, and non-diabetic patients whose blood sugar and glycated hemoglobin values cannot meet the criteria for diagnosis of T2DM, and the age is over 50 years old.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enwu Long, Master, Principal Investigator — Director of Pharmacy department
Locations (1):
- Sichuan provincial people's hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holman N, Young B, Gadsby R. Current prevalence of Type 1 and Type 2 diabetes in adults and children in the UK. Diabet Med. 2015 Sep;32(9):1119-20. doi: 10.1111/dme.12791. No abstract available. PMID 25962518
- [Background] Palermo A, Maggi D, Maurizi AR, Pozzilli P, Buzzetti R. Prevention of type 2 diabetes mellitus: is it feasible? Diabetes Metab Res Rev. 2014 Mar;30 Suppl 1:4-12. doi: 10.1002/dmrr.2513. PMID 24353270
- [Background] Lee YS, Jun HS. Anti-diabetic actions of glucagon-like peptide-1 on pancreatic beta-cells. Metabolism. 2014 Jan;63(1):9-19. doi: 10.1016/j.metabol.2013.09.010. Epub 2013 Oct 17. PMID 24140094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects ware recruited in medical clinic of Sichuan Provincial People's Hospital during July 26th 2016 to October 12th 2017.
Groups:
- Non-T2D Group: Aims to study correlationship between SNP and T2DM onset.
Period: Overall Study
Arm/Group | Sitagliptin Group | Non-T2D Group
Started | 83 | 36
Completed | 71 | 36
Not Completed | 12 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Physician Decision | 4 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin Group | Non-T2DM Group | Total
Number analyzed (Participants) | 83 | 36 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (9.7) | 60.6 (7.26) | 57.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 16 | 44
  Male | 55 | 20 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 83 | 36 | 119
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
HbA1c [Mean (Standard Deviation); unit: percentage of HbA1c] — Population: non-T2D subjects only tested HbA1c at baseline. Of the 71 patients who completed the study, 69 collected HbA1c at both baseline and study endpoint, and 2 subjects did not carry out HbA1c measurement for personal reasons.
  percentage of HbA1c
    number analyzed (Participants) | 69 | 36 | 105
    (all) | 8.26 (0.88) | 5.01 (0.67) | 7.24 (1.75)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Hemoglobin A1c (HbA1c)
Description: non-T2D subjects only tested HbA1c at baseline. Of the 71 patients who completed the study, 69 collected HbA1c at both baseline and study endpoint, and 2 subjects did not carry out HbA1c measurement for personal reasons.
Time Frame: 12 weeks later
Population: non-T2D subjects only tested HbA1c at baseline. Of the 71 patients who completed the study, 69 collected HbA1c at both baseline and study endpoint, and 2 subjects did not carry out HbA1c measurement for personal reasons.
Measure: Mean (Standard Deviation); unit: percentage of <HbA1c>
Arm/Group | Sitagliptin Group
Number analyzed (Participants) | 69
percentage of <HbA1c> | 6.78 (0.82)

2. Secondary Outcome: Types of Gene Polymorphism
Description: 24 SNPs genetic points of DPP-4, GLP-1 and GLP-1R.
Time Frame: Baseline
Population: All of the participants were detected the 24 SNPs genetic points
Measure: Number; unit: percentage of Allele frequency
Groups:
- Sitagliptin Group: Patients in this group will detect the 24 SNPs genetic points of DPP-4, GLP-1 and GLP-1R.
- Non-T2DM Group: Patients in this group also will detect the 24 SNPs genetic points of DPP-4, GLP-1 and GLP-1R.
Arm/Group | Sitagliptin Group | Non-T2DM Group
Number analyzed (Participants) | 83 | 36
percentage of Allele frequency
  rs7565794 | 40.0 | 29.2
  rs10166311 | 40.5 | 24.3
  rs2300757 | 39.2 | 25.0
  rs2302873 | 42.4 | 25.0
  rs2284872 | 42.4 | 25.0
  rs7608798 | 44.2 | 24.3
  rs2111850 | 40.5 | 25
  rs16822665 | 42.5 | 25.0

3. Secondary Outcome: Change in Blood Glucose
Description: Fasting Blood glucose, the postprandial 0.5-hour,2-hour,3-hour blood glucose were measured at baseline and at study end points, and the difference between baseline and study end points were compared.Participants in "Non-T2DM Group" were not taking Sitagliptin, so their blood glucose were not measured.
Time Frame: Basline and 12 weeks later. Fasting, 0.5h, 2h,3h after take 75g glucose orally.
Population: 71 patients complete the study
Measure: Mean (Standard Deviation); unit: mmol/l
Groups:
- Sitagliptin Group: Patients in this group will check fasting and postprandial 2-hour blood glucose
Arm/Group | Sitagliptin Group
Number analyzed (Participants) | 71
mmol/l
  ΔFasting blood glucose | -1.60 (2.29)
  Δ0.5h Glucose | -2.18 (3.11)
  Δ2h Glucose | -3.49 (4.45)
  Δ3h Glucose | -3.45 (4.36)

4. Secondary Outcome: Change in Insulin
Description: Fasting insulin, the postprandial 0.5-hour,2-hour,3-hour insulin were measured at baseline and at study end points, and the difference between baseline and study end points were compared.The changes in fasting insulin, the postprandial 0.5-hour,2-hour,3-hour insulin were compared among patients with different genotypes at baseline and at study end points.Participants in "Non-T2DM Group" were not taking Sitagliptin, so their insulin were not measured.
Time Frame: Basline and 12 weeks later. Fasting and 0.5h, 2h,3h after take 75g glucose orally.
Population: 71 patients complete the study
Measure: Mean (Standard Deviation); unit: μU/ml
Groups:
- Sitagliptin Group: To compare the baseline and endpoint insulin secretion after taking sitagliptin orally
Arm/Group | Sitagliptin Group
Number analyzed (Participants) | 71
μU/ml
  ΔFasting insulin | 0.66 (4.36)
  Δ0.5h insulin | 4.00 (8.62)
  Δ2h insulin | 8.43 (13.00)
  Δ3h insulin | 2.99 (11.77)

5. Secondary Outcome: Change in C-peptide
Description: Fasting C-peptide, the postprandial 2-hour C-peptide were measured at baseline and at study end points, and the difference between baseline and study end points were compared.The changes in fasting C-peptide, the postprandial 2-hour C-peptide were compared among patients with different genotypes at baseline and at study end points.Participants in "Non-T2DM Group" were not taking Sitagliptin, so their C-peptide were not measured.
Time Frame: Basline and 12 weeks later. Fasting and 2h after take 75g glucose orally.
Population: 71 patients complete the study
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Sitagliptin Group: Patients in this group will compare the baseline and endpoint C peptide secretion after taking sitagliptin orally
Arm/Group | Sitagliptin Group
Number analyzed (Participants) | 71
ng/ml
  ΔFasting C peptide | 0.03 (0.41)
  Δ2h C peptide | 1.11 (1.38)

ADVERSE EVENTS:
Time Frame: 3 months
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored/assessed, but no All-Cause Mortality or Serious Adverse Events observed during the study period.The dosage and administration of the drugs were not adjusted, and all adverse reactions improved after 3 days.
Arm/Group | Sitagliptin Group | Non-T2DM Group
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/36
Other Adverse Events (participants affected / at risk) | 12/71 | 0/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin Group (N=71) | Non-T2DM Group (N=36)
abdominal distension and abdominal pain 8 cases, dizziness 2 cases, constipation 2 cases (Gastrointestinal disorders) | 12 (12) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03108521/Prot_SAP_000.pdf